CLINICAL TRIAL: NCT02049294
Title: Randomized Double Blind Placebo Controlled Trial of the Steroid Sparing Effect of Xolair (Omalizumab) in Patients With Persistent Eosinophilic Bronchitis
Brief Title: Study of the Steroid Sparing Effect of Xolair (Omalizumab) in Patients With Persistent Eosinophilic Bronchitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RP 14-008
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-01

CONDITIONS: Steroid and/or Prednisone Dependent Asthma; Eosinophilic Bronchitis
Keywords: Prednisone; Eosinophils; Immunoglobin E (IgE); Asthma; Bronchitis; Inflammation; Allergy
MeSH Terms: conditions — Asthma; Bronchitis; Inflammation; Hypersensitivity | interventions — Omalizumab; anti-IgE antibodies; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omalizumab (Xolair) (Active Comparator): Dosage/frequency is dependent on body weight (kg) and baseline blood IgE level.
  Interventions: Drug: Placebo
- Placebo (Normal Saline) (Placebo Comparator): 0.9% normal saline equivalent to the dosage/frequency/duration of Omalizumab
  Interventions: Biological: Omalizumab (Xolair)

INTERVENTIONS:
Biological: Omalizumab (Xolair)
  Other Names: Anti IgE
  Arms: Placebo (Normal Saline)
Drug: Placebo
  Other Names: 0.9% normal saline
  Arms: Omalizumab (Xolair)

SUMMARY:
The purpose of this study is to investigate whether addition of Omalizumab enables a reduction in the dose of prednisone in patients with asthma and eosinophilic bronchitis.

This will be a double-blind placebo-controlled, 3-centre, randomized parallel group trial divided into two sequential study periods.

Period 1: After establishing the minimum dose of prednisone to maintain asthma control and maintain sputum eosinophils <3%, subjects will be randomized to either placebo or Omalizumab for 16 weeks (either once monthly for 4 months or every 2 weeks for 4 months).

Period 2: standardised prednisone reduction at intervals of 4-weeks until there is a clinical and eosinophilic exacerbation or bothersome steroid withdrawal effects. If patients have an exacerbation, they will be treated with prednisone. This patient will continue on Omalizumab or placebo during the entire duration of the study but not continue the phase of steroid reduction.

ELIGIBILITY:
Inclusion criteria

1. Confirmed asthma within the past 2 years (12% bronchodilator reversibility or PC20 methacholine less than 8 mg/ml)
2. ACQ ≥1.5 and sputum eos ≥3% at the time of randomization
3. On ICS (≥ 1500 mcg fluticasone propionate or equivalent) with or without additional prednisone
4. Total serum IgE ≥30 IU/L and positive allergy skin prick test
5. Age between 18 and 75 years
6. Ability to provide informed consent

Exclusion criteria

1. Current smoker or ex-smokers with greater than 20 pack years
2. Co-morbid diseases which in the investigator's opinion would make the patient unsuitable to participate in the study
3. Currently on Omalizumab or has previously been treated with Omalizumab
4. Currently on other biologic therapies (eg. Prolia)
5. Pregnancy or lactation
6. Post bronchodilator FEV1 less than 50% predicted

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-03; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with change in absolute % count of sputum eosinophil week 0 to week 12, and week 12 to week 32 | From Week 0 to Week 12 and Week 12 to week 32
Magnitude of the reduction in the dose of corticosteroid from week 12 to week 32. | From Week 12 to Week 32

SECONDARY OUTCOMES:
change in % sputum eosinophil | From Week 0 to Week 32
Blood eosinophils | From Week 0 to week 32
Forced Expired Volume in 1 second (FEV1) | From Week 0 to Week 32
Ratio of Forced Expired Volume in 1 second to Forced Vital Capacity (FEV1/VC) | From Week 0 to Week 32
Provocative concentration causing a 20% drop in FEV1 (PC20) | From Week 0 to Week 32
Asthma Control Questionnaire | From Week 0 to Week 32
Fraction of exhaled nitric oxide (FeNO) | From Week 0 to Week 32

OTHER OUTCOMES:
• Sputum eosinophilopoietic cytokines, chemokines, immunoglobulin levels, expression variation of constitutive immunoglobulin receptors. | From Week 0 to Week 12 and Week 12 to week 32
IgE antagonism and its effect on TSLP with respect to in situ eosinophilopoeisis and local eosinophil activity | From Week 0 to Week 12 and Week 12 to week 32

CONTACTS AND LOCATIONS:
Overall Officials: Parameswaran Nair, MD, PhD, Principal Investigator — McMaster University; Louis-Philippe Boulet, MD, Principal Investigator — University of Laval; Catherine Lemiere, MD, Principal Investigator — Université de Montréal; Richard Leigh, MB, Principal Investigator — University of Calgary; Delbert Dorscheid, MD, Principal Investigator — University of British Columbia
Locations (5):
- Canada (5):
  - Richard Leigh, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - McMaster University, Hamilton, Ontario
  - University of Laval, Laval, Quebec
  - University of Montreal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mukherjee M, Kjarsgaard M, Radford K, Huang C, Leigh R, Dorscheid DR, Lemiere C, Boulet LP, Waserman S, Martin J, Nair P. Omalizumab in patients with severe asthma and persistent sputum eosinophilia. Allergy Asthma Clin Immunol. 2019 Apr 3;15:21. doi: 10.1186/s13223-019-0337-2. eCollection 2019. PMID 30988677